CLINICAL TRIAL: NCT06725238
Title: The Interplay of Acute-to-Chronic Glycemic Ratio With Other Biomarkers in Diabetic Foot Ulcers: An Effect is Not Related to the Therapeutic Remedies
Brief Title: Acute-to-chronic Glycemic Ratio (ACGR) is a Marker of DFUs .
Acronym: ACGR
Status: Completed | Type: Observational
Sponsor: University of Diyala (Other)
Responsible Party: Principal Investigator, Marwan Salih Mohamad Al-Nimer, Professor of Clinical Pharmacology and Therapeutics, University of Diyala
Other Study IDs: PH130-24; University of Sulaimani (Other: College of Pharmacy)
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: Diabetes foot ulcers; Acute-to-chronic glycemic index; Leucocyte-glucose index; Triglyceride-glucose index
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I : patients presented with DFUs.: Participants who were referred to the consultant clinics at the Shar hospital were included if they had (i) a history of T2D irrespective of antidiabetic medicines or (ii) clinical and laboratory evidence of diabetic foot ulcers.
  Interventions: Other: Acute-to-chronic glycemic ratio
- Group II: patients who had T2D without DFUs: The participants have no previous history of diabetic foot ulcer or amputation. There were managed with oral anti-diabetes or occasionally with short term insulin therapy

INTERVENTIONS:
Other: Acute-to-chronic glycemic ratio — This ratio could be related to diabetic foot ulcer
  Other Names: Leucocyte glucose index; Triglyceride-glucose index
  Groups: Group I : patients presented with DFUs.

SUMMARY:
Diabetic foot ulcers (DFUs) have resulted from peripheral arterial ischemia and peripheral neuropathy that are complicated with infections and amputation of the lower extremities. Uncontrolled glycemic status and significantly higher glycosylated hemoglobin (HbA1c) are associated with DFUs. This study aimed to assess the acute-to-chronic glycemic ratio (ACGR) in type 2 diabetes (T2D) with DFUs and compare it with those without DFUs, considering the relationships of this ratio with other indices that characterized the pathogenesis of T2D. This cross-sectional study was conducted on T2D with DFUs and non-DFUs. The primary outcome is ACGR. The secondary outcomes are indices related to the anthropometric, metabolic, and hematological variables.

DETAILED DESCRIPTION:
DFUs are a macrovascular complication of diabetes mellitus resulting from peripheral artery disease and peripheral neuropathy that commonly affects the lower extremities. The DFUs are usually classified and scored according to the clinical findings. The ACGR is computed by dividing the acute (or current, or on admission in hospital) plasma glucose level by the chronic plasma glucose level calculated using the current (or on admission) HbA1c value.

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetes Clinical and laboratory diagnosis of diabetic foot ulcers Treatment with oral anti-diabetes +/- insulin

Exclusion Criteria:

History of recent systemic infections Alcohol consumption Surgical procedures within 4 weeks Pregnant or breast-feeding women; Terminal illnesses.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic participants with or without diabetic foot ulcer who were referred to the consultant clinics at the Shar hospital in Sulaymaniyah, Iraq were recruited
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Acute-to-chronic glycemic ratio | The measurement is done at the time of recruitment
  The glycemic index represents the current or acute level of fasting plasma glucose and the HbA1c, which indicates the chronic glycemic status, is elevated in DFUs. The chronic plasma glucose level could be determined by using the equation of 28.7 × HbA1c (%) - 46.7.

SECONDARY OUTCOMES:
Leucocyte-glucose index | at the time of recruitment
  Leukocyte-glucose index (LGI) combines total leukocyte and plasma glucose levels, which could serve as a prognostic biomarker of DFUs.

CONTACTS AND LOCATIONS:
Overall Officials: Rawa A Ratha, M.Sc., PhD, Principal Investigator — College of Pharmacy, University of Sulaimani, Sulaymaniyah
Locations (1):
- College of Medicine, University of Diyala, Baqubah, Diyala Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DG, Tan TW, Boulton AJM, Bus SA. Diabetic Foot Ulcers: A Review. JAMA. 2023 Jul 3;330(1):62-75. doi: 10.1001/jama.2023.10578. PMID 37395769
- See also: An article was studied the benefit of determination the stress hyperglycemia — https://doi.org/10.5603/cd.99395